Efficacy of the Female Athlete Body Project (FAB)

NCT01735994

September 4, 2019

## **Statistical Analysis**

We used linear mixed effects models with random intercept and slope, with team as the cluster level variable (N = 28), intervention as a between-subjects variable, and latent growth over the 18-month study duration as a within-subject variable. We used assessments at baseline, sixmonths, 12-months, and 18-months. Intervention effects were estimated as the between-level effects of the intervention on change at 18-months. Missing data were assumed to be missing at random, so all models use expectation-maximization likelihood estimates and included all observed data in the models. We used a maximum likelihood estimator for all models and estimated 95% confidence intervals for all model effects, unless there was evidence of variable skew, in which case we used robust maximum likelihood. Intervention effect sizes were estimated using guidelines from Fiengold, where unstandardized treatment effect (*b*) is divided by the pooled within-group *SD* at the end of treatment.